CLINICAL TRIAL: NCT06427707
Title: The Effect of Adding Either Propofol or Ketamine to Magnesium and Lidocaine Infusions As an Opioid Free Anaesthesia on Surgical Field in Patients Undergoing Nasal Surgeries. a Randomized Controlled Trial
Brief Title: The Effect of Adding Either Propofol or Ketamine to Magnesium and Lidocaine Infusions in Nasal Surgeries.
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Maher Hussien, MD, Associate Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FMASU R84/2024
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Intraoperative Bleeding
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Lidocaine; Magnesium Sulfate; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: compare the effect of; propofol- lidocaine-magnesium and ketamine- lidocaine- magnesium infusions to dexmedetomidine- lidocaine- magnesium infusion on surgical field quality in patients undergoing nasal surgeries.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group PLM (propofol-lidocaine-magnesium) (Active Comparator): intravenous infusion of propofol, lidocaine and magnesium sulfate.
  Interventions: Drug: Intravenous Infusion of propofol, lidocaine, Magnesium sulfate
- Group KLM (ketamine-lidocaine-magnesium) (Active Comparator): intravenous infusion of Ketamine, lidocaine and magnesium sulfate
  Interventions: Drug: Intravenous infusion of ketamine, lidocaine, Magnesium sulfate
- Group DLM (Dexmeditomidine-lidocaine-magnesium) (Active Comparator): Intravenous infusion of Dexmeditomidine, lidocaine and magnesium sulfate
  Interventions: Drug: Intravenous infusion of dexmedetomidine, lidocaine, Magnesium sulfate

INTERVENTIONS:
Drug: Intravenous Infusion of propofol, lidocaine, Magnesium sulfate — intravenous infusion of propofol 6-10 mg.kg-1.h-1, lidocaine (lidocaine 2% 400mg in 20 ml) bolus of 1.5 mg.kg-1 followed by infusion with a rate of 1.5 mg.kg-1.h-1 and magnesium sulfate 40 mg.kg-1 loading followed by infusion of 20 mg.kg-1.h-1. the effect of either Propofol injection, or ketamine injection or dexmeditomidine injection on intraoperative bleeding
  Arms: Group PLM (propofol-lidocaine-magnesium)
Drug: Intravenous infusion of ketamine, lidocaine, Magnesium sulfate — Patients will receive intravenous infusion of Ketamine 0.1-0.2 mg.kg-1.h-1 (intravenous infusion of propofol 6-10 mg.kg-1.h-1, lidocaine (lidocaine 2% 400mg in 20 ml) bolus of 1.5 mg.kg-1 followed by infusion with a rate of 1.5 mg.kg-1.h-1 and magnesium sulfate 40 mg.kg-1 loading followed by infusion of 20 mg.kg-1.h-1. dose of 1 mg.kg-1), lidocaine bolus of 1.5 mg.kg-1 followed by infusion with a rate of 1.5 mg.kg-1.h-1 and magnesium sulfate 40 mg.kg-1 loading followed by infusion of 20 mg.kg-1.h-1.
  Arms: Group KLM (ketamine-lidocaine-magnesium)
Drug: Intravenous infusion of dexmedetomidine, lidocaine, Magnesium sulfate — Dexmeditomidine (Precedex® 200 mcg.2ml-1) with a rate of 0.2-0.6 mcg.Kg-1.h-1. lidocaine bolus of 1.5 mg.kg-1 followed by infusion with a rate of 1.5 mg.kg-1.h-1 and magnesium sulfate 40 mg.kg-1 loading followed by infusion of 20 mg.kg-1.h-1
  Other Names: Precedex
  Arms: Group DLM (Dexmeditomidine-lidocaine-magnesium)

SUMMARY:
Nasal surgeries are common day case procedures. Although surgical complications are rare, bleeding decreases surgical field visibility and may cause vascular, orbital or intracranial complications in addition to failure of procedure. So, it is crucial to maintain hypotensive anaesthesia to optimize the surgical field.

DETAILED DESCRIPTION:
In this study the investigators compare the effect of; propofol- lidocaine-magnesium and ketamine- lidocaine- magnesium infusions to dexmedetomidine- lidocaine- magnesium infusion on surgical field quality, intraoperative haemodynamics, surgical time, recovery time, sedation score, time to first rescue analgesic and incidence of PONV in patients undergoing nasal surgeries

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II,
* scheduled for elective nasal surgery

Exclusion Criteria:

* Patients with uncontrolled hypertension.
* Patients with cardiac disease.
* Patients with renal, hepatic or cerebral insufficiency.
* Patients with coagulopathy or receiving drugs influencing blood coagulation.
* Anaemia, haemoglobinopathies or polycythemia.
* Pregnancy.
* Patients with known sensitivity to any of the study drug.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
surgical field using the average category scale (ACS). | During the operation
  Degree of surgical field bleeding

SECONDARY OUTCOMES:
sedation using Ramsy sedation score | First hour postoperative
  Degree of sedation using Ramsy sedation score

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Cairo Governorate, Egypt